CLINICAL TRIAL: NCT06031545
Title: An Exploratory Study of Perioperative Venous Access in Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20230718072255619
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Catheter Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Not possible because of the material and characteristics of the catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long peripheral venous catheters (Experimental): In the test group used LPCs during the perioperative period in obese patients
  Interventions: Other: Long peripheral venous catheters for use
- Midline catheters (Other): In the control group used LPCs during the perioperative period in obese patients
  Interventions: Other: Midline catheter

INTERVENTIONS:
Other: Long peripheral venous catheters for use — Long peripheral venous catheters for use during the perioperative period in obese patients
  Arms: Long peripheral venous catheters
Other: Midline catheter — Midline catheters for use during the perioperative period in obese patients
  Arms: Midline catheters

SUMMARY:
This study is intended to explore the application effect of long peripheral intravenous catheters(LPCs) and midline catheters(MCs) in the perioperative period of obese patients, aiming at providing the scientific basis for the optimal perioperative venous access for the obese patients.

DETAILED DESCRIPTION:
This study is intended to explore the application effect of long peripheral intravenous catheters(LPCs) and midline catheters(MCs) in the perioperative period of obese patients; at the same time, the LPCs will be used as the control group and the MCs as the experimental group, to compare whether the application of LPCs in the perioperative period of obese patients is not inferior to that of the MCs; the comprehensive comparison of the effect of the clinical application and the evaluation of the health economics, aiming at providing the scientific basis for the optimal perioperative venous access for the obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI ≥ 30kg/m2) who are to undergo surgery.
* Expected length of hospitalisation within 2 weeks.
* Conscious and able to communicate normally.

Exclusion Criteria:

* It is expected that perioperative medications will need to be infused via a central venous catheter (e.g. total parenteral nutrition TPN);
* Patients with an indwelling central venous catheter on admission

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Catheter-related complication rate | during catheter indwelling,an average of 2 weeks
  The proportion of patients with complications as a proportion of the total number of cases

SECONDARY OUTCOMES:
Catheter retention days | during catheter indwelling,an average of 2 weeks
  Number of days from the day of catheter placement to the day of extubation
Completion rate of treatment via one catheter | during catheter indwelling,an average of 2 weeks
  Number of patient cases in which all infusion treatments were completed via one catheter/total number of patient cases

CONTACTS AND LOCATIONS:
Overall Officials: Linfang Zhao, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Linfang Zhao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
You can email if you need to

REFERENCES:
- [Background] Pan XF, Wang L, Pan A. Epidemiology and determinants of obesity in China. Lancet Diabetes Endocrinol. 2021 Jun;9(6):373-392. doi: 10.1016/S2213-8587(21)00045-0. PMID 34022156
- [Background] Kivimaki M, Strandberg T, Pentti J, Nyberg ST, Frank P, Jokela M, Ervasti J, Suominen SB, Vahtera J, Sipila PN, Lindbohm JV, Ferrie JE. Body-mass index and risk of obesity-related complex multimorbidity: an observational multicohort study. Lancet Diabetes Endocrinol. 2022 Apr;10(4):253-263. doi: 10.1016/S2213-8587(22)00033-X. Epub 2022 Mar 4. PMID 35248171
- [Background] Zheng Y, Manson JE, Yuan C, Liang MH, Grodstein F, Stampfer MJ, Willett WC, Hu FB. Associations of Weight Gain From Early to Middle Adulthood With Major Health Outcomes Later in Life. JAMA. 2017 Jul 18;318(3):255-269. doi: 10.1001/jama.2017.7092. PMID 28719691
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Juvin P, Blarel A, Bruno F, Desmonts JM. Is peripheral line placement more difficult in obese than in lean patients? Anesth Analg. 2003 Apr;96(4):1218. doi: 10.1213/01.ANE.0000050570.85195.29. PMID 12651688
- [Background] Keogh S, Shelverton C, Flynn J, Mihala G, Mathew S, Davies KM, Marsh N, Rickard CM. Implementation and evaluation of short peripheral intravenous catheter flushing guidelines: a stepped wedge cluster randomised trial. BMC Med. 2020 Sep 30;18(1):252. doi: 10.1186/s12916-020-01728-1. PMID 32993628
- [Background] Shokoohi H, Boniface K, McCarthy M, Khedir Al-tiae T, Sattarian M, Ding R, Liu YT, Pourmand A, Schoenfeld E, Scott J, Shesser R, Yadav K. Ultrasound-guided peripheral intravenous access program is associated with a marked reduction in central venous catheter use in noncritically ill emergency department patients. Ann Emerg Med. 2013 Feb;61(2):198-203. doi: 10.1016/j.annemergmed.2012.09.016. Epub 2012 Nov 7. PMID 23141920
- [Background] Chopra V, Flanders SA, Saint S, Woller SC, O'Grady NP, Safdar N, Trerotola SO, Saran R, Moureau N, Wiseman S, Pittiruti M, Akl EA, Lee AY, Courey A, Swaminathan L, LeDonne J, Becker C, Krein SL, Bernstein SJ; Michigan Appropriateness Guide for Intravenouse Catheters (MAGIC) Panel. The Michigan Appropriateness Guide for Intravenous Catheters (MAGIC): Results From a Multispecialty Panel Using the RAND/UCLA Appropriateness Method. Ann Intern Med. 2015 Sep 15;163(6 Suppl):S1-40. doi: 10.7326/M15-0744. PMID 26369828
- [Background] Nielsen EB, Antonsen L, Mensel C, Milandt N, Dalgaard LS, Illum BS, Arildsen H, Juhl-Olsen P. The efficacy of midline catheters-a prospective, randomized, active-controlled study. Int J Infect Dis. 2021 Jan;102:220-225. doi: 10.1016/j.ijid.2020.10.053. Epub 2020 Oct 28. PMID 33129962
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Derived] Zhao L, Yang X, Liu C, Yu W, Cao X, Li X, Wang J, Zhuang Y. Comparative safety and efficacy of midline catheters versus long peripheral catheters in patients undergoing bariatric surgery: a randomised controlled trial. Sci Rep. 2025 Aug 20;15(1):30534. doi: 10.1038/s41598-025-12551-0. PMID 40835653